CLINICAL TRIAL: NCT05961891
Title: The Use of Composite Bone and Nail Bed Graft Combined With Cutaneous Flaps for Reconstruction of Finger Tip Amputations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hassan Abdellatif Hamed, Resident-plastic department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-07-02MS
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Finger Tip Amputations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Finger Tip Amputations (Experimental): Patients with Finger Tip Amputations
  Interventions: Procedure: The Use of Composite Bone and Nail Bed Graft Combined With Cutaneous Flaps for Reconstruction of Finger Tip Amputations

INTERVENTIONS:
Procedure: The Use of Composite Bone and Nail Bed Graft Combined With Cutaneous Flaps for Reconstruction of Finger Tip Amputations — 1. The amputated finger tip is cleaned and a composite graft including the nail bed and bone of distal phalanx is taken from the amputated part.
  2. The bone of the amputated part is fixed to the remaining stump of the distal phalanx with an axial 21gauge needle or by a K-wire (0.8 mm).
  3. The nail bed graft is sutured with 6-0 vicryl to the remaining nail bed.
  4. A local or regional cutaneous flap is used to cover the volar aspect and tip of the distal phalanx bone e.g. V-Y advancement flap, thenar flap or cross finger flap .The flap should protrude beyond the tip, providing extra skin which is recontoured to a rounded tip.
  5. The nail plate is inserted in the nail fold to prevent the formation of synechiae between the nail fold and the injured nail bed.
  6. The finger is immobilized for two weeks in a below elbow dorsal slab.
  7. Patients are followed up for 3 months. Postoperative complications and their management will be recorded.

SUMMARY:
Fingertip injuries are among the most common hand injuries regardless of age, as the fingertip is a prominent and frequently used part of the hand. However, no consensus yet exists regarding the ideal reconstruction of fingertip injuries with nail bed defects, and its reconstructive methods are limited.

Allen has classified fingertip amputations into four types. Type I injuries involve only the pulp of the finger. Type II includes pulp and nail loss. Type III has partial terminal phalanx loss and corresponding pulp and nail loss. Finally, type IV involves the lunule of the nail, pulp, nail, and partial loss of the terminal phalanx.

Fingertip amputations through the proximal half of the nail-bed are challenging as the remaining nail-bed has inadequate length for satisfactory nail growth. Replantation at this level gives a good functional and cosmetic results but is technically demanding, requires microsurgical skills and adequate facilities and is not always possible.When replantation is not possible, the use of a local advancement palmar flap preserves digital length and the remaining nail bed.

However, when the amputation is through the proximal third of the nail, this technique leaves very little nail bed and nail deformities are common.To avoid these deformities, complete ablation of the nail bed and germinal matrix with closure by a palmar advancement flap, or by shortening, are usually carried out. Unfortunately, these treatments often fail to satisfy the patient's desire to retain his or her nail.

When replantation is not feasible, the technique of advancing a palmar V-Y flap and applying the nail bed retrieved from the amputated part to the dorsum of the flap provides an alternative means of restoring nail bed length. So the technique of using composite bone and nail bed graft from the amputated part with a local or regional cutaneous flaps may be an option for treatment of fresh fingertip amputation to restore the shape and preserve the length of the fingertip especially in circumstances when microsurgical replantation is not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Any level of finger tip amputations through the nail bed and distal phalanx with preserved amputated part.

Exclusion Criteria:

* Crushed part of amputated segment.
* Patients with peripheral vascular disease.
* Diabetic patient.
* Pateint over 65 or under 5 years of age.
* Patient refusal.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Fingertip length | 1 year
  Fingertip length is estimated in Centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allen MJ. Conservative management of finger tip injuries in adults. Hand. 1980 Oct;12(3):257-65. doi: 10.1016/s0072-968x(80)80049-0. PMID 7002744
- [Background] Brown RE, Zook EG, Russell RC. Fingertip reconstruction with flaps and nail bed grafts. J Hand Surg Am. 1999 Mar;24(2):345-51. doi: 10.1053/jhsu.1999.0345. PMID 10194021
- [Background] Celik N, Wei FC, Lin CH, Cheng MH, Chen HC, Jeng SF, Kuo YR. Technique and strategy in anterolateral thigh perforator flap surgery, based on an analysis of 15 complete and partial failures in 439 cases. Plast Reconstr Surg. 2002 Jun;109(7):2211-6; discussion 2217-8. doi: 10.1097/00006534-200206000-00005. PMID 12045538
- [Background] Cheung K, Hatchell A, Thoma A. Approach to traumatic hand injuries for primary care physicians. Can Fam Physician. 2013 Jun;59(6):614-8. PMID 23766041